CLINICAL TRIAL: NCT06156956
Title: Fecal Microbiota Transplantation to Eradicate Antibiotic-resistance Bacteria From the Gastrointestinal Tract of Patients at High Risk of Infection and/or to Cut Off the Spread of Bacteria With Dangerous Mechanisms of Antibiotic Resistance
Brief Title: Fecal Microbiota Transplantation (FMT) to Decolonize Antibiotic - Resistant Bacteria (ARB) - New Protocol
Acronym: STOP-ARB2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Human Biome Institute S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI/2023/01/STOP-ARB2
Record Dates: First submitted 2023-10-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Drug Resistance, Bacterial; Antimicrobial Drug Resistance
Keywords: Antibiotic-resistant bacteria decolonization; Gastrointestinal tract colonization; Eradication procedure; Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Single group, open label, observational study with intervention (Fecal Microbiota Transplantation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Antibiotics pre-treatment on days 1-5 and a bowel cleansing on day 6. Days 7-14 are dedicated to active eradication treatment with FMT. First dose on day 7 and second dose in days 9-14 (1/6 of full dose every day).
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation in capsules or suspension obtained from healthy unrelated donor introduced two times per treatment:
  for capsules - FMT administration: day 7 (full dose) and days from 9 to 14 (prolonged intake regimen)
  for suspension - FMT administration: day 7 and day 14
  Other Names: MBiotix HBI

SUMMARY:
The aim of the study is to assess the safety and efficacy of new protocol fecal microbiota transplantation (FMT) in the eradication of antibiotic resistant bacteria, including those featuring of resistance to new generation antibiotics.

This study should answer the following research questions:

1. Will new treatment protocol and fully anaerobic FMT be effective in decolonization of ARB?
2. Will FMT improve the prognosis and quality of life in patients at high risk of ARB infection?

DETAILED DESCRIPTION:
Fecal microbiota transplantation (FMT) was shown to be very efficient in treatment of relapsed and refractory Clostridium difficile infection and became a standard treatment. The investigators company produces and uses FMT not only in case of Clostridioides difficile colitis, but also in case of gut colonization with antibiotic-resistant bacteria and other indications as a clinical studies under Bioethical Committee approval. Company's flagship program to decolonize ARB is based on assumption that physiological gut flora may outcompete the pathogenic bacteria similarly as in case of Clostridium difficile and lead to loss of colonization.

Patients colonized with ARB are characterized by poor diversity of gut microbiome (dysbiosis), which makes them vulnerable to further infections. In case of gut mucosa injury and severe immune suppression, these colonizing bacteria may cause severe systemic infections.

During this interventional prospective, single arm, observational study, the investigators collect the information about the safety and effectiveness of FMT in gut decolonization with antibiotic-resistance bacteria (ARB) using their new treatment protocol and own full-spectrum, full-richness, full-viability anaerobic FMT.

The project protocol is based on the intervention (fecal microbiota transplantation; FMT) in capsules (or colonoscopy if per os route is not possible) applied twice - on day 7th after procedure initiation and between day 9-14 within extended period, low dose (1/6th every day) application. All patient are premedicated with non-absorbable antibiotics on days 1-5 and a bowel cleansing on day 6 from the screening. After the end of the eradication procedure, the patient proceeds to the follow-up assessment stage and is observed up to 360 days with longitudinal samples collection.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 6 months
2. Population of patients colonized with antibiotic-resistant bacteria, as follows:

   1. strains of antibiotic-resistant bacteria that exhibit resistance mechanisms to carbapenems (MBL+: NDM+, VIM+ or others), KPC+, OXA-48+ or confirmed resistance to carbapenems without a specific genetic mechanism
   2. strains of Enterobacteriaceae resistant to beta lactams and other antibiotics in the case of multi-drug resistance (e.g. in the ESBL resistance mechanism and others) of the types including Escherichia, Enterobacter, Klebsiella, strains of P. aeruginosa, A. baumannii (together included in, among others, the ESKAPE group)
   3. Gram (+) enterococci E. faecalis or E. faecium or other bacteria resistant to vancomycin (VRE), linezolid and strains of S. aureus resistant to methicillin (MRSA) or vancomycin
   4. other multidrug-resistant or drug-resistant strains with threatening clinical resistance mechanisms or in patients vulnerable to infection with a particular pathogen
3. Absolute neutrophil count in the peripheral blood up to 3 days before FMT > 500/ul (in the case of tandem multiple FMTs, in patients with an expected decrease in neutrophil values, the test should be repeated before each FMT when the timeframe between FMTs is longer than 3 days, and in patients without an expected decrease in the value of neutrophils below 500 cells/ul peripheral blood counts are valid for 28 days)
4. Signing of the informed consent for participation in the study.

Exclusion Criteria:

1. Inability to obtain informed consent and lack of consent
2. Blood neutrophil count <500/uL on the day of fecal microbiota transplantation or expected decrease to the mentioned number within 2 consecutive days
3. Active infection requiring intensive antimicrobial treatment on FMT day or the first 7 days after FMT in immunocompetent patients (without immunosuppression or immunodeficiency)
4. Clinical signs of mucositis 7 days prior to FMT
5. Contraindications to FMT via upper and lower gastrointestinal tract (e.g. perforation of the digestive tract, rectal atresia, discontinuity of the digestive tract and others)
6. Severe food allergy with the anaphylaxis history

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication of gut colonizing antibiotic-resistant bacteria | Baseline, 30, 60, 90, 180, 360 days after the end of eradication
  The effectiveness of the therapy is assessed by means of rectal swabs and/or stool cultures after 30, 60, 90, 180 and 360 days (i.e. after a month, two, three and six) from the end of the eradication procedure

SECONDARY OUTCOMES:
Increase in the diversity of the recipients' gut microbiota | from pre-treatment to 360 days after-treatment
  Assesment of microbiome changes after treatment through a multi-omic analysis

OTHER OUTCOMES:
Infections-oriented safety profile assessment | During 3 months form FMT
  Number of adverse events (AE) regarding infectious complications after FMT

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Bilinski, MD, PhD, Principal Investigator — Human Biome Institute S.A.
Locations (5):
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Klinika Gastroenterologii i Hepatologii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Klinika Pediatrii, Hematologii i Onkologii, Gdansk
  - WOJEWÓDZKI SZPITAL ZESPOLONY W KIELCACH, Klinika Chorób Zakaźnych, Kielce
  - WIM-PIB: Klinika Chorób Infekcyjnych i Alergologii, Klinika Gastroenterologii i Chorób Wewnętrznych, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rokkas T, Gisbert JP, Gasbarrini A, Hold GL, Tilg H, Malfertheiner P, Megraud F, O'Morain C. A network meta-analysis of randomized controlled trials exploring the role of fecal microbiota transplantation in recurrent Clostridium difficile infection. United European Gastroenterol J. 2019 Oct;7(8):1051-1063. doi: 10.1177/2050640619854587. Epub 2019 May 27. PMID 31662862
- [Background] Maier L, Pruteanu M, Kuhn M, Zeller G, Telzerow A, Anderson EE, Brochado AR, Fernandez KC, Dose H, Mori H, Patil KR, Bork P, Typas A. Extensive impact of non-antibiotic drugs on human gut bacteria. Nature. 2018 Mar 29;555(7698):623-628. doi: 10.1038/nature25979. Epub 2018 Mar 19. PMID 29555994
- [Background] Chung H, Pamp SJ, Hill JA, Surana NK, Edelman SM, Troy EB, Reading NC, Villablanca EJ, Wang S, Mora JR, Umesaki Y, Mathis D, Benoist C, Relman DA, Kasper DL. Gut immune maturation depends on colonization with a host-specific microbiota. Cell. 2012 Jun 22;149(7):1578-93. doi: 10.1016/j.cell.2012.04.037. PMID 22726443
- [Background] Buffie CG, Pamer EG. Microbiota-mediated colonization resistance against intestinal pathogens. Nat Rev Immunol. 2013 Nov;13(11):790-801. doi: 10.1038/nri3535. Epub 2013 Oct 7. PMID 24096337
- [Background] Diehl GE, Longman RS, Zhang JX, Breart B, Galan C, Cuesta A, Schwab SR, Littman DR. Microbiota restricts trafficking of bacteria to mesenteric lymph nodes by CX(3)CR1(hi) cells. Nature. 2013 Feb 7;494(7435):116-20. doi: 10.1038/nature11809. Epub 2013 Jan 13. PMID 23334413
- [Background] Bilinski J, Grzesiowski P, Sorensen N, Madry K, Muszynski J, Robak K, Wroblewska M, Dzieciatkowski T, Dulny G, Dwilewicz-Trojaczek J, Wiktor-Jedrzejczak W, Basak GW. Fecal Microbiota Transplantation in Patients With Blood Disorders Inhibits Gut Colonization With Antibiotic-Resistant Bacteria: Results of a Prospective, Single-Center Study. Clin Infect Dis. 2017 Aug 1;65(3):364-370. doi: 10.1093/cid/cix252. PMID 28369341
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Kronman MP, Zerr DM, Qin X, Englund J, Cornell C, Sanders JE, Myers J, Rayar J, Berry JE, Adler AL, Weissman SJ. Intestinal decontamination of multidrug-resistant Klebsiella pneumoniae after recurrent infections in an immunocompromised host. Diagn Microbiol Infect Dis. 2014 Sep;80(1):87-9. doi: 10.1016/j.diagmicrobio.2014.06.006. Epub 2014 Jun 21. PMID 25041704